CLINICAL TRIAL: NCT02385448
Title: A Prospective, Randomized Controlled Trial Comparing the Use of Dienogest and Combined Oral Contraceptive Pills (Microgynon) to Reduce the Risk of Recurrence of Endometriotic Cyst After Conservative Surgery
Brief Title: Comparing the Use of Dienogest and Combined Oral Contraceptive Pills (Microgynon) to Reduce the Risk of Recurrence of Endometriotic Cyst After Conservative Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 14-097
Record Dates: First submitted 2015-02-12; First posted 2015-03-11 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-03

CONDITIONS: Endometriosis
Keywords: dienogest; combined oral contraceptive pills; endometriosis
MeSH Terms: conditions — Endometriosis | interventions — dienogest; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dienogest (Experimental)
  Interventions: Drug: Dienogest
- Combined oral contraceptive pills (Active Comparator)
  Interventions: Drug: Microgynon

INTERVENTIONS:
Drug: Dienogest — The dienogest group will receive dienogest 2mg daily for 24 months postoperatively
  Other Names: Visanne
  Arms: Dienogest
Drug: Microgynon — The combined oral contraceptive pills group will be given cyclical Microgynon for 24 months.
  Arms: Combined oral contraceptive pills

SUMMARY:
The purpose of the study is to compare the recurrence of endometriotic cyst in patients taking Dienogest or Microgynon after conservative surgery.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Older than the age of legal consent (i.e. 18 years old)
* Sonographic diagnosis of ovarian endometrioma with diameter at least 4cm on 2 separate scans at least 6 weeks apart
* No contraindication to use of progesterone or combined oral contraceptive pills
* Not attempting to conceive either at the time of study entry or for at least 2 years after surgery
* Willing and able to participate after the study has been explained

Exclusion Criteria:

* Operative findings not suggestive of endometriotic cyst
* Contraindications to progestogens or oral contraceptive pills
* Unwillingness to tolerate menstrual irregularity
* Planning pregnancy within 2 years of study
* Cannot understand English, Cantonese or Putonghua

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence of ovarian endometrioma | 2 years
  Time to recurrence by sonography (months)
Recurrence of ovarian endometrioma | 2 years
  Size of recurrent endometrioma on sonography (mean diameter in centimeters)

SECONDARY OUTCOMES:
Side effects | 2 years
  Days of irregular bleeding
Symptoms of endometriosis | 2 years
  Pain by visual analog score
Need for additional analgesics | 2 years
  Types of analgesics used

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K.Y. Ko, MBBS, MRCOG, Principal Investigator — The University of Hong Kong, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong